CLINICAL TRIAL: NCT04943146
Title: An Assessment of Aspirin Plus Prednisone Treatment for Euthyroid Women With Thyroid Autoimmunity Undergoing In Vitro Fertilization
Brief Title: An Assessment of Aspirin Plus Prednisone Treatment for Euthyroid Women With Thyroid Autoimmunity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo Women & Children's Hospital (Other); People's Hospital of Jinhua (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-0062
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-03

CONDITIONS: Thyroid Diseases
Keywords: Prednisolone; Assisted reproductive technology; Aspirin; thyroid diseases
MeSH Terms: conditions — Thyroid Diseases | interventions — Prednisone; Aspirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control group
- P+A group: aspirin: tablet 100mg qd 2-5weeks prednisone: tablet 10mg qd 2-5weeks
  Interventions: Drug: Prednisone 10 MG+aspirin 100MG

INTERVENTIONS:
Drug: Prednisone 10 MG+aspirin 100MG — Discontinue medication based on early pregnancy outcome
  Groups: P+A group

SUMMARY:
Thyroid autoimmunity(TAI) per se have adverse effect on pregnancy outcomes，and aspirin and prednisone were used frequently in antithyroid antibodies(ATA) positive infertile women in clinical practice, but the impact of these medicines is still controversial. Therefore, aim of the study was to investigate whether or not the treatment of prednisone in addition to aspirin was capable of improving reproductive outcomes in euthyroid infertile women.

DETAILED DESCRIPTION:
A multicenter retrospective study performed during the period of 2017 to 2020 and euthyroid infertile women positive for anti-thyroperoxidase antibody (TPOAb) and/or thyroglobulin antibody (TgAb) alone with thyroid stimulating hormone 0.35-4.0mIU/L undergoing first in vitro fertilization and embryo transfer(IVF-ET) cycle were recruited in our study.Data analysis was performed using the Statistics Package for Social Sciences.In the end, the value of prednisone plus aspirin treatment was investigated to make a big contribution on clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Both TPOAb and TgAb in all the subjects were measured before ART procedure
2. Thyroid stimulating hormone (TSH) level ranged from 0.35-4.0mIU/L
3. Women underwent first embryo transfer without previous IVF history.

Exclusion Criteria:

1. Abnormal thyroid function test
2. Women with known autoimmune diseases or clinical presentations of autoimmune disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — we investigate pregnant women
Study Population: Both TPOAb and TgAb in all the subjects were measured before ART procedure, and their thyroid stimulating hormone (TSH) level ranged from 0.35-4.0mIU/L and also they all underwent first embryo transfer without previous IVF history.
Sampling Method: Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 3 mouths
  Clinical pregnancy was defined as the existence of a viable embryo within an intrauterine gestational sac

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - People's Hospital of Jinhua, Jinhua, Zhejiang
  - Ningbo Women and Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
uncertainty